CLINICAL TRIAL: NCT04167735
Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application
Brief Title: Assessment of Novel Sound Changing Principles in Hearing Instruments to Determine Their Application - 2019_33
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2019_33
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Aid without Reverberation Canceller (no_RevC) (Active Comparator): Hearing Aid without Reverberation Canceller (RevC)
  Interventions: Device: Hearing Aid without Reverberation Canceller (RevC).
- : Hearing Aid Reverberation Canceller enabled (RevC_1) (Experimental): Hearing Aid Reverberation Canceller enabled (RevC_1)
  Interventions: Device: Hearing Aid Reverberation Canceller enabled (RevC_1)

INTERVENTIONS:
Device: Hearing Aid without Reverberation Canceller (RevC). — Each participant will be fitted with the 2 different Sound Changing principles on the same hearing aid, saved to 2 manual programs (ensures exact same hearing loss compensation for each intervention). Reverberation Canceller principle is a sound processing algorithm to remove reverberation from a speech signal to improve the speech intelligibility and comfort. The active comparator condition is without Reverberation Canceller principle enabled.
  Arms: Hearing Aid without Reverberation Canceller (no_RevC)
Device: Hearing Aid Reverberation Canceller enabled (RevC_1) — Each participant will be fitted with the 2 different Sound Changing principles on the same hearing aid, saved to 2 manual programs (ensures exact same hearing loss compensation for each intervention). Reverberation Canceller principle is a sound processing algorithm to remove reverberation from a speech signal to improve the speech intelligibility and comfort. The experimental condition applies the Reverberation Canceller and is predicted to provide a benefit in reverberant room simulations.
  Arms: : Hearing Aid Reverberation Canceller enabled (RevC_1)

SUMMARY:
Participants will complete a listening task in a simulated reverberant environment. Participants are seated and instructed to look at a fixation cross while a sentence is played. Sentences are varied with respect to their speech rate. While listening to the sentences participant's pupil dilation is measured by means of pupillometry which is a non-invasive physiological measurement. Participants are asked to repeat back the sentences loud. At fixed intervals, subjective ratings are collected by asking participants to move an on-screen slider using a game controller. Two hearing aid programs will be compared, one intended for speech perception in quiet and the other to reduce reverberation in reverberant environments. The study is designed as factorial, with 2 speech rates, 2 room simulations and 2 hearing aid programs. The same conditions will be re-tested once after a minimum of one day. A pilot study will determine appropriate speech rates by applying a different factorial, with 4 speech rates, 2 room simulations and 1 hearing aid program. Participants complete all conditions (within-subjects) in one experimental sessions that lasts around 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature
* Mild-Moderate/Severe (N2-N4) hearing loss

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Changes in Event-related-pupil-dilations (ERPDs) | 4 weeks
  Pupil dilations will be recorded from the participant during the performance of the auditory tasks. Analyses will be carried out relative to the pre-trial baseline (measured one second prior to the onset of the stimulus), in order to account for differences in baseline physiological activity. It is planned to analyze event-related-pupil-dilations.

SECONDARY OUTCOMES:
Oldenburg sentence test | 4 weeks
  1. Words recalled correctly: words repeated back by participants are logged and the percentage of words recalled correctly calculated.
subjective rating | 4 weeks
  Subjective ratings: using a game controller, participants rate the difficulty of the sentences and listening effort on a visual analog scale. The scale is continuous and ranges from minimal to maximal difficulty/effort. The position of the cursor on the scale is then used to calculate a percentage from 0-100% difficulty/effort.

OTHER OUTCOMES:
Non-verbal Trail Making Test A & B | 1 week
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The data, serving as an outcome measure, are time-to-complete the set in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No